CLINICAL TRIAL: NCT05110482
Title: Carbetocin Versus Syntocinon for Prevention of Postpartum Hemorrhage in Cardiac Patients With Stenotic Valvular Heart Disease Undergoing Caesarean Section
Brief Title: Carbetocin Versus Syntocinon for Prevention of Postpartum Hemorrhage in Cardiac Patients Undergoing Caesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, Assistant professor of anesthiology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD-247-2020
Record Dates: First submitted 2021-09-28; First posted 2021-11-08 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Adverse Effect of Oxytocic Drugs
MeSH Terms: interventions — Oxytocin; carbetocin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- syntocinon group (Active Comparator): in this group :5 mL syringe containing a bolus of 1 IU of oxytocin and infusion syringe which will be prepared with a 50 mL syringe containing 0.4 IU/mL of oxytocin and infusion rate of 7.5 IU/h will be administrated to the patient after delivery of the fetus shoulder, Additional bolus syringes will be prepared for use as rescue boluses if needed " which will be 5 ml syringe containing 3 IU of oxytocin
  Interventions: Drug: Syntocinon
- carbetocin group (Active Comparator): in this group :5 mL syringe containing a bolus of 100 mcg of carbetocin and infusion syringe " which will be prepared with a 50 mL syringe containing normal saline will be administrated for the patient after delivery of the fetus shoulder. Additional bolus syringes will be prepared for use as rescue boluses if needed which will be 5 ml syringe containing 100 mcg of carbetocin
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Syntocinon — uterotonic drugs
  Arms: syntocinon group
Drug: Carbetocin — uterotonic drug
  Arms: carbetocin group

SUMMARY:
Postpartum hemorrhage (PPH) is the primary cause of nearly one quarter of all maternal deaths globally. Management of uterine tone after delivery involves giving a prophylactic uterotonic and the use of controlled cord traction to facilitate delivery of the placenta and minimize blood loss. Syntocinon and carbetocin are the most commonly used drugs ,During caesarean delivery of stenotic valvular disease patient, the anesthesiologist have an important question: what is the best drug used for prevention of PPH with minimal hemodynamic effect regarding Systemic vascular resistance (SVR), Cardiac out put (COP),Heart rate ( HR), blood pressure? As uterotonic drugs may cause severe hypotension, decrease in SVR and COP that may not be tolerated by these patients .this thesis aims to compare between syntocinon and carbetocin regarding their effect on cardiac output and systemic vascular resistance using cardiometry in cardiac patients with stenotic lesions during caesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female single tone >38 weeks
* Age :18-45 years old.
* patient with ASA III
* Cardiac patients ( mild and moderate mitral stenosis-aortic stenosis valve disease )

Exclusion Criteria:

* Other cardiac conditions (valve regurge, cardiomyopathy, heart failure,severe mitral stenosis, severe aortic stenosis, severe pulmonary hypertension)
* Pregnancy hypertensive disorders (eclampsia,preeclampsia)
* Abnormal placental attachment (accrete,percreta,increta)
* Patients with bleeding disorders
* patient with high risk of postpartum haemorrhage

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females presented for caesarean delivery
Enrollment: 38 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | intraoperative
  Average Cardiac output after study drug administration

SECONDARY OUTCOMES:
systemic vascular resistance | intraoperative
  Systemic vascular resistance every 2 minute till end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine CAIRO UNIVERISTY, Cairo, Egypt